CLINICAL TRIAL: NCT01562496
Title: The ParkCycle Study: Effects of Aerobic Exercise on Cognitive and Adaptive Plasticity in Parkinson's Disease
Brief Title: The ParkCycle Study: Aerobic Exercise in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL38116.091.11
Record Dates: First submitted 2012-03-19; First posted 2012-03-23 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Neuroprotective; Intensive exercise
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Twente patients will perform Aerobic exercise 3 times a week for at least 30 min
  Interventions: Behavioral: Exercise
- Control (No Intervention): Fifteen patients will be listed as a control group and will be instructed to continue their previous level of activity throughout the study

INTERVENTIONS:
Behavioral: Exercise — six-months long exercise intervention on a stationary virtual reality bike, 3-5 times a week, each session lasting 30-45 minutes at a target heart rate (60-85% heart rate reserve).
  Arms: Exercise

SUMMARY:
The primary goal of this study is to determine the neuroprotective qualities of long-term, in home, exercise therapy program in human PD patients. It is hypothesized that an exercise intervention might delay the onset of levo-dopa therapy (i.e. evidence for neuroprotection). The first part involves a pilot-study in which the feasibility of the intervention and outcome measures will be tested.

DETAILED DESCRIPTION:
Neuroprotective therapy (i.e. therapy that slows the disease process) is an unmet medical need in Parkinson's disease (PD). Animal studies have shown that 'intensive' exercise improves motor function and may have neuroprotective properties. The promising animal results have not been translated to patients with PD so far. This is a two-cluster randomised control trial in which twenty patients (10 at each site) will undergo a 6-month exercise intervention on a stationary virtual reality bike and twenty patients (10 at each site)will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease according to the UK Queen Square Brain Bank Criteria
* Hoehn & Yahr disease stages I-II
* Age between 30 and 75 years
* Having insufficient physical activity according to the ACSM guideline for adults, 50-64 years old with a chronic condition
* Untreated with anti-parkinsonian medication or receiving medication, for less than two years, medication-responsive without fluctuations.

Exclusion Criteria:

* Unclear diagnosis with Red Flags
* Advanced problems in cognitive functioning: Mini Mental State Examination (MMSE)19 score < 24
* Serious co-morbidity: neurological or orthopedic disorder that severely affects movement; known by specialist or medical practitioner
* Pulmonary diseases; known by specialist or medical practitioner
* Stroke
* High risk of cardiovascular complications:

  * Hypertension (systole >150 and diastole > 100)
  * Diabetes Mellitus; known by specialist or medical practitioner
  * Cardiac valve defect (especially aortic valve stenosis); known by specialist or medical practitioner
  * Cardiac rhythm disorder; known by specialist or medical practitioner
  * Heart failure; known by specialist or medical practitioner
* Use of ß-blockers
* Not able to complete American (for Cleveland site) or Dutch questionnaires (for the Nijmegen site)
* Daily institutionalized care
* Contra-indications for fMRI:

  * Pregnancy
  * Metallic implants or electronic devices
  * Previous seizure
  * Claustrophobia
  * Not able to keep the head still for longer period, i.e. due to severe head tremor

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Trails A and B task | every month for 6-7 months
  this test requires subjects to connect numbers on a screen from 1 to 25 (part A) and to connect numbers to letters. This neuropsychological test has already been proven to be sensitive to frontal lobe damage (e.g. Boll 1981) and has been recognised as an outcome for executive function in PD21. This test is performed using an online system called i-COMET that allows subject to complete the task weekly at home. Subjects have to login at the i-COMET website (https://i-comet.com) with a username and password that is provided to them by the research team.

SECONDARY OUTCOMES:
UPDRS | baseline and after 6 months follow-up (FU)
Cognitive tests | baseline and after 6 months FU
  MMSE and SCOPA-org
Kinetics tests | baseline and after 6 months FU
  Timed Up and Go Test (iTUG) and a postural sway test, , as an objective measure for balance and mobility Finger tap test as a measure for bradykinesia and a pegboard test as a measure for complex motor function
questionaires | baseline and after 6 months FU
  The PDQ-39 is a PD specific questionnaire including 39 items concerning quality of life. Other non-motor features such as mood and sleep are respectively measured using the HADS and SCOPA-Sleep.
maximal exercise test | baseline and after 6 months FU
  to determine training load and subject fitness
feasibility parameters | after 6 months (termination of intervention)
  Compliance based on the number of completed exercise sessions and the amount of time that patients exercised at their target heart rate.
neuroplasticity | baseline and after 6 months FU
  1. Volumetric brain changes: cerebral grey and white matter will be analyzed using Vox-Based Morphometry, a validated and fully automated technique for computational analysis of differences in global and local grey and/or white matter volume.
  2. Resting state brain perfusion: functional coupling between strial subregions and the cerebral cortex will be analyzed using multiple regression analyses on resting state functional MRI data.

CONTACTS AND LOCATIONS:
Overall Officials: Bas Bloem, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Cleveland clinic, Cleveland, Ohio, United States
- UMC St Radboud, Nijmegen, Netherlands

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886